CLINICAL TRIAL: NCT03416088
Title: The Influence of Daily Activities on Retinal Microcirculation in Normal Adults
Brief Title: Influence of Daily Activities on Retinal Microcirculation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jiannan Huang (Other)
Responsible Party: Sponsor-Investigator, Jiannan Huang, Director, Shanghai Eye Disease Prevention and Treatment Center
Organization: Shanghai Eye Disease Prevention and Treatment Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: YFZX2017001
Record Dates: First submitted 2018-01-17; First posted 2018-01-30 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Retinal Microcirculation Disorder
Keywords: Beverage consumption; Reading; Body motion; Retinal microcirculation; Optical coherence tomography angiography; Magnetic resonance imaging

STUDY DESIGN:
Intervention Model Description: 1. Influence of beverage consumption Participants drink coffee, red wine, Baijiu (Chinese liquor), grape juice, and water respectively on three mornings with one-week washout. Each period lasts 2 hours. An additional test with SipSparkTM Probiotics (facilitates ethanol degradation) was taken 0.5 hour prior to Baijiu consumption. OCTA and MRI scanning are taken every 30 minutes, and venous blood is collected.
  2. Influence of daily reading 30 participants read paper books, play video games with mobile phones, and non-read respectively on three mornings interval with one-week washout. OCTA and MRI scanning are taken every 2 hours for a total of 8 hours.
  3. Influence of body motion Exercise: 30 participants are enrolled. Participants undergo to jogging for 10 minutes, 30 minutes, and 1 hour respectively on three mornings with a 3-day washout. Body postural changes: 30 participants are enrolled. OCTA and MRI scanning are taken before and after jogging or body postural changes.
Who Masked: Outcomes Assessor
Masking Description: Data analyzers are blind to the participants classification
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Beverage consumption (Experimental): Drink 300ml red wine (alcohol concentration:12.5%), 300ml coffee (caffeine concentration 72 mg), 300 ml Baijiu (Chinese liquor, alcohol concentration:12.5%) , SipSparkTM Probiotics (facilitates ethanol degradation) was taken 0.5 hour prior to Baijiu consumption, or 300ml water.
  Interventions: Behavioral: Beverage consumption
- Daily reading (Experimental): Reading paper books, playing video games with mobile phones, or non-reading.
  Interventions: Behavioral: Daily reading
- Body motion (Experimental): Exercise and body postural changes.
  Interventions: Behavioral: Body motion

INTERVENTIONS:
Behavioral: Beverage consumption — The participants drink 300ml wine (alcohol concentration:12.5%)or 300ml coffee (caffeine concentration 72 mg), or water.
  Arms: Beverage consumption
Behavioral: Daily reading — Reading paper books, playing video games with mobile phones, or non-reading for 8 hours.
  Arms: Daily reading
Behavioral: Body motion — Exercise or body postural changes
  Arms: Body motion

SUMMARY:
The daily behaviors such as drinking coffee, wine, reading, exercise and body postural changes may have influence on the function or morphology of the retinal microcirculation in healthy people.A recent study found that the fingertips microvascular bed constricted obviously after the intake of a cup of coffee with caffeine, it significantly reduced blood flow to the fingers; Long reading of electronic products can induce significant dry eye symptoms, affect visual quality, and cause asthenopia. Microcirculation is critical for regulating vascular resistance and blood flow in organs. Fundus blood vessels is the only visible microvascular in vivo, its morphology and function changes not only associated with eye disease, but also with cardiovascular and cerebrovascular diseases. Optical coherence tomography angiography (OCTA) is a new technique which could acquire blood flow information in a non-invasive way without the use of dye. Magnetic resonance imaging (MRI) can quantitatively evaluation of cerebral blood flow and retina-choroid blood flow using the noninvasive arterial spin labeling technique in a large field of view (FOV) without depth limitations.The study tried to detect the influence of daily behaviors such as drinking coffee, red wine, reading , exercise, etc. on the retinal microcirculation with OCTA and MRI, and provide reference for health behaviors.

ELIGIBILITY:
Inclusion Criteria

1. Healthy adults
2. The age range was from 18 to 35 years old
3. Without another eye disease besides ametropia
4. The spherical equivalent is equal or above minus 3.00 diopters
5. No smoking or drinking
6. Average daily caffeine consumption no more than 1 cup of coffee
7. No diabetes, hypertension, heart disease, liver or kidney dysfunction
8. No medication taken recently

Exclusion Criteria

1. Mental disorders such as depression and anxiety
2. Intellectual disabilities
3. Female in menstruation, gestation period, perinatal period or lactation period
4. Unable to cooperate with eye examinations and test procedures
5. Heart disease, hypertension, diabetes, liver and kidney dysfunction and other chronic diseases
6. Patients with fever, acute infectious diseases
7. Other conditions that are not suitable for drinking alcohol or coffee, such as allergic to alcohol or coffee

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Vessel diameter index (VDI) | 3 weeks
  VDI is calculated using both the vessel area map and the skeletonized vessel map, to yield the averaged vessel caliber.
Vessel area density (VAD) | 3 weeks
  VAD is calculated as a unit-less ratio of the total image area occupied by the vasculature to the total image area in the binary vessel maps.
Flow impairment region (FIR) | 3 weeks
  FIZ: calculated by summing all 'no-flow' pixels up.
Retina-choroid blood flow | 3 weeks
  Blood flow for the entire retinal thickness were determined as a function of the distance from the optic nerve head, where the blood flow was measured at the peaks of the projection profiles. An region of interest outlining the posterior retina with a size of 0.7 to 0.8 mm across the retina-choroid thickness in the parafoveal region was used to obtain the blood flow signal time courses and averaged the values.
Cerebral blood flow (CBF) | 3 weeks
  The frontal lobe was selected as the region of interest (ROI) to measure and average the changes in CBF

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Eye Disease Prevention & Treatment Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data because of personal privacy.

REFERENCES:
- [Background] Malerba S, Turati F, Galeone C, Pelucchi C, Verga F, La Vecchia C, Tavani A. A meta-analysis of prospective studies of coffee consumption and mortality for all causes, cancers and cardiovascular diseases. Eur J Epidemiol. 2013 Jul;28(7):527-39. doi: 10.1007/s10654-013-9834-7. Epub 2013 Aug 11. PMID 23934579
- [Background] Ronksley PE, Brien SE, Turner BJ, Mukamal KJ, Ghali WA. Association of alcohol consumption with selected cardiovascular disease outcomes: a systematic review and meta-analysis. BMJ. 2011 Feb 22;342:d671. doi: 10.1136/bmj.d671. PMID 21343207
- [Background] Lawrenson JG, Hull CC, Downie LE. The effect of blue-light blocking spectacle lenses on visual performance, macular health and the sleep-wake cycle: a systematic review of the literature. Ophthalmic Physiol Opt. 2017 Nov;37(6):644-654. doi: 10.1111/opo.12406. PMID 29044670
- [Result] Karti O, Zengin MO, Kerci SG, Ayhan Z, Kusbeci T. ACUTE EFFECT OF CAFFEINE ON MACULAR MICROCIRCULATION IN HEALTHY SUBJECTS: An Optical Coherence Tomography Angiography Study. Retina. 2019 May;39(5):964-971. doi: 10.1097/IAE.0000000000002058. PMID 29401177
- [Result] Luksch A, Resch H, Weigert G, Sacu S, Schmetterer L, Garhofer G. Acute effects of intravenously administered ethanol on retinal vessel diameters and flicker induced vasodilatation in healthy volunteers. Microvasc Res. 2009 Sep;78(2):224-9. doi: 10.1016/j.mvr.2009.06.001. Epub 2009 Jun 10. PMID 19523476
- [Result] Strang NM, Claus ED, Ramchandani VA, Graff-Guerrero A, Boileau I, Hendershot CS. Dose-dependent effects of intravenous alcohol administration on cerebral blood flow in young adults. Psychopharmacology (Berl). 2015 Feb;232(4):733-44. doi: 10.1007/s00213-014-3706-z. Epub 2014 Aug 12. PMID 25110231
- [Result] Kojima S, Sugiyama T, Kojima M, Azuma I I, Ito S. Effect of the consumption of ethanol on the microcirculation of the human optic nerve head in the acute phase. Jpn J Ophthalmol. 2000 May;44(3):318-9. doi: 10.1016/s0021-5155(00)00158-1. PMID 10913661
- [Result] Molnar F, Frank CC. Determining the causes of postural hypotension. Can Fam Physician. 2018 Jan;64(1):40. No abstract available. PMID 29358250